CLINICAL TRIAL: NCT05290961
Title: Drug Response in Patient-derived Organoids Models of Advanced or Recurrent Ovarian Cancer, an Exploratory Research
Brief Title: The Culture of Advanced or Recurrent Ovarian Cancer Organoids and Drug Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Other Study IDs: CQGOG0202
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian Neoplasms; Organoids; Drug Screening
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Ovarian cancer tissues were cut into 1-3 mm3 pieces. Two random pieces were snap frozen and stored at -80℃ for DNA isolation, two random pieces were fixed in formalin for histopathological analysis and immunohistochemistry, and the remainder was processed for organoids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — The study is an observational trial, which don't have any intervention.

SUMMARY:
Most ovarian cancer will relapse after standard therapy. Patients with recurrent ovarian cancer are resistant to platinum. Due to the high heterogeneity between ovarian cancer, individual precise therapy is of great importance. The study will establish ovarian cancer organoids, whose original tissues from the patients with advanced or recurrent ovarian cancer, their tumors cannot be excised completely. The organoids will be identified at the histopathological level and gene level for evaluating the consistency with the original tumor tissue. The drug's sensitivity and specificity are detected through the organoids model. Compared with the clinical efficiency of the actual drug regimen, the efficacy of the organoid drug screening model can be assessed. The aim is to construct a precise drug screening platform for advanced and recurrent ovarian cancer patients and innovate drug research and development.

DETAILED DESCRIPTION:
This trial is a single-arm and prospective observational study. The subjects are the advanced or recurrent ovarian cancer patients, who are planned to undergo surgery, but the neoplastic lesions can't be excised thoroughly. They voluntarily participate in the study and sign an informed consent form. General information will be collected, including name, age, address and contact information. Comprehensive physical examination will be performed. Ovarian cancer tumor markers and imaging examinations (gastroenterostomy, ultrasound / CT / MRI or PET / CT) should be taken within 4 weeks before treatment. Histopathological and genetic characteristics were analyzed in organoids and paired primary tumors to confirm whether organoids faithfully recapitulated the original tumor tissues. The sensitivity and specificity of first-line and second-line drugs from NCCN guidelines will be detected on the organoids. Ovarian cancer (CA125、HE4、CEA、CA-199) markers will be tested within one week. After the treatment period of 3 and 6 months, the short-term efficacy will be evaluated according to the efficacy evaluation standard of solid tumor (Recist1.1) (the window period is 4 weeks). Biochemical indexes, adverse reactions, and prognosis (PFS, OS) will be followed. Compared with the efficacy of the actual clinical regimen, the potency of organoid as a drug screening model will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and signed informed consent;
2. The tumour cannot be excised thoroughly by surgery;
3. ECOG score ≤ 2;
4. Expected survival >6 months;
5. Blood routine test: Hb≥70g/L、WBC≥3.5×109/ L 、ANC≥1.5×109/L、PLT≥80×109/L;
6. Both serum ALT and serum AST ≤ 2 × ULN； blood creatinine ≤ 1.5 × ULN;
7. Unpregnant women (negative HCG) received contraception in the study;
8. Good compliance is judged by researchers.

Exclusion Criteria:

1. Active or the uncontrol serious infections;
2. Patients with liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need antiviral treatment;
3. A history of immune deficiency, including HIV positive or other acquired congenital immune deficiency diseases;
4. Chronic renal insufficiency and renal failure;
5. Myocardial infarction, severe arrhythmia and congestive heart failure (≥ grade 2 according to NYHA classification);
6. Autoimmune diseases, including systemic lupus erythematosus;
7. Patients take drugs that damage liver and kidney function for other complications, such as tuberculosis;
8. Patients cannot understand the experimental contents and refuse to sign the informed consent form;
9. Other concomitant serious diseases harm the health of patients or interfere with the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with advanced or recurrent ovarian cancer, who are planned to undergo surgery, but the tumour cannot be excised thoroughly. They voluntarily participate in the study and sign an informed consent form.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 2 years
  Progression-free survival means the duration from enrollment to disease progression or death.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival means the duration from enrollment to death due to any cause. The last follow-up time is calculated as the death time for subjects who lost follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
These individual participant data (IPD) involves patients' informed consent and our technical confidentiality.

REFERENCES:
- [Background] Tuveson D, Clevers H. Cancer modeling meets human organoid technology. Science. 2019 Jun 7;364(6444):952-955. doi: 10.1126/science.aaw6985. PMID 31171691
- [Background] Sachs N, Clevers H. Organoid cultures for the analysis of cancer phenotypes. Curr Opin Genet Dev. 2014 Feb;24:68-73. doi: 10.1016/j.gde.2013.11.012. Epub 2013 Dec 31. PMID 24657539
- [Background] Chen Z, Fillmore CM, Hammerman PS, Kim CF, Wong KK. Non-small-cell lung cancers: a heterogeneous set of diseases. Nat Rev Cancer. 2014 Aug;14(8):535-46. doi: 10.1038/nrc3775. PMID 25056707
- [Background] Bertotti A, Migliardi G, Galimi F, Sassi F, Torti D, Isella C, Cora D, Di Nicolantonio F, Buscarino M, Petti C, Ribero D, Russolillo N, Muratore A, Massucco P, Pisacane A, Molinaro L, Valtorta E, Sartore-Bianchi A, Risio M, Capussotti L, Gambacorta M, Siena S, Medico E, Sapino A, Marsoni S, Comoglio PM, Bardelli A, Trusolino L. A molecularly annotated platform of patient-derived xenografts ("xenopatients") identifies HER2 as an effective therapeutic target in cetuximab-resistant colorectal cancer. Cancer Discov. 2011 Nov;1(6):508-23. doi: 10.1158/2159-8290.CD-11-0109. Epub 2011 Sep 2. PMID 22586653
- [Background] Zhao X, Liu Z, Yu L, Zhang Y, Baxter P, Voicu H, Gurusiddappa S, Luan J, Su JM, Leung HC, Li XN. Global gene expression profiling confirms the molecular fidelity of primary tumor-based orthotopic xenograft mouse models of medulloblastoma. Neuro Oncol. 2012 May;14(5):574-83. doi: 10.1093/neuonc/nos061. Epub 2012 Mar 29. PMID 22459127
- [Background] Bergamaschi A, Hjortland GO, Triulzi T, Sorlie T, Johnsen H, Ree AH, Russnes HG, Tronnes S, Maelandsmo GM, Fodstad O, Borresen-Dale AL, Engebraaten O. Molecular profiling and characterization of luminal-like and basal-like in vivo breast cancer xenograft models. Mol Oncol. 2009 Dec;3(5-6):469-82. doi: 10.1016/j.molonc.2009.07.003. Epub 2009 Aug 4. PMID 19713161
- [Background] Sato T, Vries RG, Snippert HJ, van de Wetering M, Barker N, Stange DE, van Es JH, Abo A, Kujala P, Peters PJ, Clevers H. Single Lgr5 stem cells build crypt-villus structures in vitro without a mesenchymal niche. Nature. 2009 May 14;459(7244):262-5. doi: 10.1038/nature07935. Epub 2009 Mar 29. PMID 19329995
- [Background] Brancati G, Treutlein B, Camp JG. Resolving Neurodevelopmental and Vision Disorders Using Organoid Single-Cell Multi-omics. Neuron. 2020 Sep 23;107(6):1000-1013. doi: 10.1016/j.neuron.2020.09.001. PMID 32970995
- [Background] Rossi G, Manfrin A, Lutolf MP. Progress and potential in organoid research. Nat Rev Genet. 2018 Nov;19(11):671-687. doi: 10.1038/s41576-018-0051-9. PMID 30228295
- [Background] Heo I, Dutta D, Schaefer DA, Iakobachvili N, Artegiani B, Sachs N, Boonekamp KE, Bowden G, Hendrickx APA, Willems RJL, Peters PJ, Riggs MW, O'Connor R, Clevers H. Modelling Cryptosporidium infection in human small intestinal and lung organoids. Nat Microbiol. 2018 Jul;3(7):814-823. doi: 10.1038/s41564-018-0177-8. Epub 2018 Jun 25. PMID 29946163
- [Background] Sato T, Stange DE, Ferrante M, Vries RG, Van Es JH, Van den Brink S, Van Houdt WJ, Pronk A, Van Gorp J, Siersema PD, Clevers H. Long-term expansion of epithelial organoids from human colon, adenoma, adenocarcinoma, and Barrett's epithelium. Gastroenterology. 2011 Nov;141(5):1762-72. doi: 10.1053/j.gastro.2011.07.050. Epub 2011 Sep 2. PMID 21889923
- [Background] Boj SF, Hwang CI, Baker LA, Chio II, Engle DD, Corbo V, Jager M, Ponz-Sarvise M, Tiriac H, Spector MS, Gracanin A, Oni T, Yu KH, van Boxtel R, Huch M, Rivera KD, Wilson JP, Feigin ME, Ohlund D, Handly-Santana A, Ardito-Abraham CM, Ludwig M, Elyada E, Alagesan B, Biffi G, Yordanov GN, Delcuze B, Creighton B, Wright K, Park Y, Morsink FH, Molenaar IQ, Borel Rinkes IH, Cuppen E, Hao Y, Jin Y, Nijman IJ, Iacobuzio-Donahue C, Leach SD, Pappin DJ, Hammell M, Klimstra DS, Basturk O, Hruban RH, Offerhaus GJ, Vries RG, Clevers H, Tuveson DA. Organoid models of human and mouse ductal pancreatic cancer. Cell. 2015 Jan 15;160(1-2):324-38. doi: 10.1016/j.cell.2014.12.021. Epub 2014 Dec 31. PMID 25557080
- [Background] Ganesh K, Wu C, O'Rourke KP, Szeglin BC, Zheng Y, Sauve CG, Adileh M, Wasserman I, Marco MR, Kim AS, Shady M, Sanchez-Vega F, Karthaus WR, Won HH, Choi SH, Pelossof R, Barlas A, Ntiamoah P, Pappou E, Elghouayel A, Strong JS, Chen CT, Harris JW, Weiser MR, Nash GM, Guillem JG, Wei IH, Kolesnick RN, Veeraraghavan H, Ortiz EJ, Petkovska I, Cercek A, Manova-Todorova KO, Saltz LB, Lavery JA, DeMatteo RP, Massague J, Paty PB, Yaeger R, Chen X, Patil S, Clevers H, Berger MF, Lowe SW, Shia J, Romesser PB, Dow LE, Garcia-Aguilar J, Sawyers CL, Smith JJ. A rectal cancer organoid platform to study individual responses to chemoradiation. Nat Med. 2019 Oct;25(10):1607-1614. doi: 10.1038/s41591-019-0584-2. Epub 2019 Oct 7. PMID 31591597
- [Background] Gao D, Vela I, Sboner A, Iaquinta PJ, Karthaus WR, Gopalan A, Dowling C, Wanjala JN, Undvall EA, Arora VK, Wongvipat J, Kossai M, Ramazanoglu S, Barboza LP, Di W, Cao Z, Zhang QF, Sirota I, Ran L, MacDonald TY, Beltran H, Mosquera JM, Touijer KA, Scardino PT, Laudone VP, Curtis KR, Rathkopf DE, Morris MJ, Danila DC, Slovin SF, Solomon SB, Eastham JA, Chi P, Carver B, Rubin MA, Scher HI, Clevers H, Sawyers CL, Chen Y. Organoid cultures derived from patients with advanced prostate cancer. Cell. 2014 Sep 25;159(1):176-187. doi: 10.1016/j.cell.2014.08.016. Epub 2014 Sep 4. PMID 25201530